CLINICAL TRIAL: NCT01809938
Title: Gastric Emptying of Tea With Milk, Compared With Tea Without Milk. Does Milk Delay Gastric Emptying?
Brief Title: Does Adding Milk to Tea Delay Gastric Emptying?
Acronym: GETEAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Sam Hillyard, Anaesthetic Registrar, Guy's and St Thomas' NHS Foundation Trust
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: STH01
Record Dates: First submitted 2013-03-07; First posted 2013-03-13 (Estimated); Results first posted 2013-10-30 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2013-11

CONDITIONS: Gastric Emptying
Keywords: Gastrointestinal tract emptying; Pre-operative fasting; Ultrasound; Paracetamol Absorption
MeSH Terms: interventions — Tea; Milk

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Black Tea (Active Comparator)
  Interventions: Other: Black tea
- Tea with Milk (Active Comparator)
  Interventions: Other: Tea with milk

INTERVENTIONS:
Other: Black tea — 300ml of tea without milk
  Arms: Black Tea
Other: Tea with milk — 250ml of black tea with 50ml of full fat milk
  Arms: Tea with Milk

SUMMARY:
Most pre-operative fasting regimes dictate that if there is any milk added to tea or coffee, the preoperative fasting time should be extended from 2 to 6 hours. The purpose of this study is to demonstrate whether there is really a delay in gastric emptying time associated with the inclusion of milk in a cup of tea.

DETAILED DESCRIPTION:
This was a randomised controlled crossover study conducted in ten healthy volunteers. The paracetamol absorption technique and real-time ultrasound measurement of the cross-sectional area (CSA) of the gastric antrum were used to assess gastric emptying following ingestion of 300ml of black tea or 300ml of tea with milk (250ml black tea plus 50ml of full fat milk)

Each participant took part in both arms of the trial, drinking black tea and tea with milk, the order of which was determined by a computerised random number generator and concealed from the investigators by opaque brown paper envelopes.

In each arm of the study the procedure was as follows. The subject sat in a semi-reclined position at a 45 angle, a 16g intravenous cannula was sited in an upper limb and baseline blood samples taken. The initial cross-sectional area of the gastric antrum was then measured by ultrasound.

The investigating anaesthetist then left the room, the subject opened their randomisation envelope and drank, as directed, either 300ml of black tea or 300ml of tea with milk (250ml black tea plus 50ml of full fat milk) over 3 minutes, followed by 1.5 g of dispersible paracetamol dissolved in 30ml of water.

Blood samples were taken every 10 minutes for the first hour, then every 30 minutes until 150 minutes had elapsed. Paracetamol concentrations in each sample were measured using an enzymatic assay. Time to peak concentration (tmax) was thus determined.

The CSA of the gastric antrum was measured by ultrasound in real-time (RUS) at baseline, every ten minutes for 60 minutes and then at 30-minute intervals for 150 minutes. Antral CSA was plotted against time and gastric emptying expressed as half-time to gastric emptying (T½). This was defined as the time from baseline to the time the gastric antrum returns to half the maximal value.

The primary outcome was tmax. Previous studies have shown mean or median tmax values for paracetamol to vary from 25 to 60 minutes following ingestion of clear fluids, with standard deviation up to 38 minutes. In this study we considered that a delay of gastric emptying of under 60 minutes would not be clinically important; and that we would be able to declare that the two regimes were equivalent if the (two sided) 95% confidence interval for the mean difference in tmax, between black tea and tea with milk included only times less than 60 minutes. Using these assumptions and taking (pessimistically) a correlation between repeated measurements of 0.0, power analysis determined nine participants would be required (with 90% power) to show equivalence.

A 95% confidence interval for the mean difference in tmax that lay entirely within 60 minutes of no effect would confirm the hypothesis that tea with milk was clinically equivalent to black tea.

ELIGIBILITY:
Inclusion Criteria:

* Healthy non-pregnant volunteers

Exclusion Criteria:

* medical conditions with a predisposition to delayed gastric emptying (e.g. diabetes or gastric disease)
* ingestion of paracetamol within the previous 24 hours
* ingestion of solids or non-clear liquids in the previous six hours
* ingestion of clear liquids in the previous two hours.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2011-11; Primary Completion 2012-01 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Geraldine O'Sullivan, Principal Investigator — St Thomas' Hospital, Guy's & St Thomas' NHS Foundation Trust
Locations (1):
- St Thomas' Hospital, London, United Kingdom

REFERENCES:
- [Background] Smith I, Kranke P, Murat I, Smith A, O'Sullivan G, Soreide E, Spies C, in't Veld B; European Society of Anaesthesiology. Perioperative fasting in adults and children: guidelines from the European Society of Anaesthesiology. Eur J Anaesthesiol. 2011 Aug;28(8):556-69. doi: 10.1097/EJA.0b013e3283495ba1. PMID 21712716
- [Background] Wong CA, Loffredi M, Ganchiff JN, Zhao J, Wang Z, Avram MJ. Gastric emptying of water in term pregnancy. Anesthesiology. 2002 Jun;96(6):1395-400. doi: 10.1097/00000542-200206000-00019. PMID 12170052
- [Background] Darwiche G, Almer LO, Bjorgell O, Cederholm C, Nilsson P. Measurement of gastric emptying by standardized real-time ultrasonography in healthy subjects and diabetic patients. J Ultrasound Med. 1999 Oct;18(10):673-82. doi: 10.7863/jum.1999.18.10.673. PMID 10511299

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place from november 2011 until january 2012 at St Thomas' Hospital, London
Groups:
- Black Tea First, Then Tea With Milk: Effects on gastric emptying of Black tea (300ml of tea without milk) were assessed then after a period of not less than 24 hours the effects of Tea with Milk (250mls of tea with 50mls of full fat millk) were assessed
- Tea With Milk First Then Black Tea: Effects on gastric emptying of Tea with Milk (250mls of tea with 50mls of full fat millk) were assessed then after a period of not less than 24 hours the effects of Black tea (300ml of tea without milk) were assessed.
Period: First Intervention (170 Minutes)
Arm/Group | Black Tea First, Then Tea With Milk | Tea With Milk First Then Black Tea
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0
Period: Washout (Not Less Than 24 Hours)
Arm/Group | Black Tea First, Then Tea With Milk | Tea With Milk First Then Black Tea
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0
Period: Second Intervention (170 Minutes)
Arm/Group | Black Tea First, Then Tea With Milk | Tea With Milk First Then Black Tea
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The the total number of participants was 10, each participant completed both arms of the trial.
Groups:
- Entire Study Population: Includes all participants in this crossover trial
Arm/Group | Entire Study Population
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Region of Enrollment [Number; unit: participants]
  United Kingdom | 10

OUTCOME MEASURES:

1. Primary Outcome: Tmax
Description: tmax = the time taken to reach peak paracetamol concentration. The blood samples were analysed for the level of paracetamol, from which the time taken to reach peak paracetamol concentration was subsequently calculated. Blood samples were taken at the same time points as the ultrasound measurements.
Time Frame: Blood samples taken every 10 minutes for 1 hour and then 30 minute intervals until 150 minutes had elapsed. Each participant spent approximately 3 hours for each arm of the trial separated by no less than 24 hours
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- Black Tea: Black tea : 300ml of tea without milk
- Tea With Milk: Tea with milk : 250ml of black tea with 50ml of full fat milk
Arm/Group | Black Tea | Tea With Milk
Number analyzed (Participants) | 10 | 10
minutes | 38 (17.6) | 30 (23.9)

2. Secondary Outcome: T½
Description: T½ = time from baseline to the time the cross-sectional surface area (CSA) of the gastric antrum, measured using realtime ultrasound, returned to half the maximal value (CSA½max ). CSA ½ max calculated as below:
  CSA½max = CSAmax - [(CSAmax - CSAbaseline)/2]
Time Frame: Measurments taken every 10 minutes for 1 hour and then 30 minute intervals until 150 minutes had elapsed. Each participant spent approximately 3 hours for each arm of the trial separated by no less than 24 hours.
Population: It was difficult to visualise under ultrasound the gastric antrum in one patient after they drank both black tea and tea with milk, so they were exlcuded from final analysis of the US data only.
Measure: Geometric Mean (95% Confidence Interval); unit: minutes
Arm/Group | Black Tea | Tea With Milk
Number analyzed (Participants) | 9 | 9
minutes | 22.7 [12.7 to 40.9] | 23.6 [13.5 to 41]

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Entire Study Population
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes